CLINICAL TRIAL: NCT05285059
Title: Implicit Learning in Epileptic Children
Acronym: IMPLICIT
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_1190
Record Dates: First submitted 2022-03-07; First posted 2022-03-17 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Epilepsy
Keywords: Epilepsy,; children,; implicit learning
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: 8- to 14-years-old children with epilepsy
  Interventions: Behavioral: ASRT task
- Control: 8- to 14-years-old children without neurological, psychiatric, or developmental impairments
  Interventions: Behavioral: ASRT task

INTERVENTIONS:
Behavioral: ASRT task — The ASRT (Alternating Serial Reaction Time) task is a computerized behavioral task measuring implicit learning. This task consists of 20 series of trials lasting 2 minutes each.
  In each trial, a stimulus is displayed on the screen in one of the four possible predefined locations. The participant must press a button to indicate the position of the stimulus on the screen. Response content and response time are recorded.
  At the end of every trial, the participant can take a break and resume the task whenever ready. The task lasts about 45 to 50 minutes.

SUMMARY:
Epileptic children suffer from impairments in various learning and memory tasks. Yet, no study investigated implicit learning in epileptic children. Implicit learning is not only underlying motor skills acquisition, but also social and cognitive ones. Because acquisition of new skills is optimal during childhood, the study of implicit learning mechanism in children is of major importance. The present study will be the first to explore implicit learning mechanisms in children with epilepsy. Implicit learning mechanisms can be preserved or altered.

ELIGIBILITY:
Inclusion Criteria:

* For Patient group only: Children with epilepsy
* For Control group only: Children without neurological, psychiatric or developmental impairments
* For both groups: Parent or tutors agreement
* For both groups: Affiliated to French social security

Exclusion Criteria:

* Neurological impairments unrelated to epilepsy
* Psychiatric impairments unrelated to epilepsy
* Developmental impairments unrelated to epilepsy

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This study focuses on children with epilepsy.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-03-21 (Actual); Primary Completion 2026-03-21 (Estimated); Study Completion 2026-03-21 (Estimated)

PRIMARY OUTCOMES:
Response time | The day of the inclusion
  Response time (in milliseconds) recorded during the ASRT task
Response accuracy recorded during the ASRT task | The day of the inclusion
  Response accuracy (percentage of correct answers)

CONTACTS AND LOCATIONS:
Overall Officials: Marcastel Agathe, PhD, Principal Investigator — Service d'Epileptologie Clinique, des Troubles du sommeil et de Neurologie fonctionnelle de l'enfant - Hôpital Femme Mère Enfant
Locations (3):
- France (3):
  - Agathe Marcastel, PhD, Bron
  - Dezso Nemeth, Bron
  - Service d'Epileptologie Clinique, des Troubles du sommeil et de Neurologie fonctionnelle de l'enfant, à Hôpital Femme Mère et Enfant,, Bron

IPD SHARING:
Plan to Share IPD: No